CLINICAL TRIAL: NCT01411722
Title: Electrical Activity of the Diaphragm in Mechanically Ventilated Patients During the Weaning Period
Brief Title: Electrical Activity of the Diaphragm During the Weaning Period
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Marco Ranieri, MD Professor, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EADIWEANIG299
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Respiratory Insufficiency
Keywords: Electrical Activity of Diaphragm; Weaning outcome; NAVA
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EADIWEANING (Other): Patients mechanically ventilated for more than 48 hours during the weaning process.
  Interventions: Device: Neurally adjust ventilatory assist (NAVA) and a nasogastric tube to measure the electrical activity of the diaphragm (EAdi catheter)

INTERVENTIONS:
Device: Neurally adjust ventilatory assist (NAVA) and a nasogastric tube to measure the electrical activity of the diaphragm (EAdi catheter) — Nava is a new ventilatory mode which delivers pressure in proportion of the the Electrical activity of the diaphragm (EAdi), a reflection of the neural respiratory output. EAdi will be obtained through a nasogastric tube with a multiple array of electrodes placed at its distal end. Correct positioning of the EAdi catheter is assured by means of a specific function of the ventilator (''EAdi catheter positioning''). The EAdi signal is processed according to the American Thoracic Society (ATS) recommendations and filtered by algorithms designed to provide the highest possible signal-to-noise ratio

SUMMARY:
The study aims to assess 1) the electrical activity of the diaphragm in mechanically ventilated patients during weaning from mechanical ventilation. 2) Whether the electrical activity of the diaphragm may predict the weaning outcome

DETAILED DESCRIPTION:
Optimization of the time to liberate the patient from mechanical ventilation should be balanced between the risks associated with failed extubation and those related to prolonged mechanical ventilation. Weaning failure is associated with major complications. Even when weaning protocols and clinical predictors have been used to improve the weaning outcome, there is still a significant proportion of patients who fail to breath spontaneously with significant risks of pneumonia, prolonged mechanical ventilation and increased morbidity and mortality rate. Electrical activity of the diaphragm, a mirror of the respiratory drive and now available on an ICU ventilator may help to predict in a more accurate way the weaning outcome. The patients will be ventilated in NAVA with the titration method (1). As soon as patients passed successfully a daily screening EAdi will be measured during a spontaneous breathing trial.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years and mechanically ventilated for >= 48 h.
* In the resolving stage of the disease which brought to mechanical ventilation.
* Pao2/Fio2 ratio >150 on positive end-expiratory pressure (PEEP) <=8 cm H2O.
* Sedation discontinued for a minimum of 24 hrs
* Analgesia provided solely with morphine at a dosage of less or equal to 0.01 mg/kg/hr.
* Patient fully alert and cooperative.
* Intact respiratory drive evaluated with Glasgow Coma Scale >=10.

Exclusion Criteria:

* The attending physician refuses to allow enrolment
* The patient refuses informed consent
* Hemodynamic instability despite adequate filling (i.e. need for continuous infusion of epinephrine or vasopressin, or dopamine or dobutamine > 5 mcg/kg/min or norepinephrine > 0.1 mcg/kg/min to maintain systolic arterial blood pressure > 90 mmHg)
* No collaborative Patient
* Coagulation or platelets disorders
* neuromuscular disease
* phrenic nerve damage/diaphragm paralysis
* contraindication to exchange naso-gastric tube
* History of heart or lung transplantation
* Presence or suspicion of a central nervous system disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-09; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Electrical activity of the diaphragm as a predictor of weaning outcome | 48 hours

SECONDARY OUTCOMES:
Comparison of electrical activity of the diaphragm as a predictor versus other predictors | 48 hours
Evaluation of respiratory parameters during the weaning process | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Ranieri, Co.so Bramante 88, Torino, Italy